CLINICAL TRIAL: NCT03921372
Title: Optic Nerve Head Blood Flow Regulation During Isometric Exercise in Patients With Normal Tension Glaucoma
Brief Title: Isometric Exercise in NTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Principal Investigator, Matthias Bolz, Prof., Augenabteilung Allgemeines Krankenhaus Linz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IsometricProtocol2
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Mean Blur Ratio
Keywords: Normal tension glaucoma
MeSH Terms: conditions — Low Tension Glaucoma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Tension Glaucoma (NTG) (Experimental): Patients with diagnosed NTG
  Interventions: Diagnostic Test: Isometric exercise
- Healthy Control Subjects (Experimental): Subjects with no sign of glaucoma, Age and sex matched
  Interventions: Diagnostic Test: Isometric exercise

INTERVENTIONS:
Diagnostic Test: Isometric exercise — Squatting for 5 minutes

SUMMARY:
Glaucoma is the second leading cause of blindness worldwide. Literature shows increasing evidence that dysfunction of ocular microcirculation in the optic nerve influences the progression of glaucoma. It has been shown that flicker light-induced vasodilatation of retinal veins is diminished in patients with glaucoma. Also previous studies indicate that the blood flow autoregulation is impaired in patients with glaucoma. Therefor the ocular perfusion pressure can not be maintained stable during changes of the systemic arterial blood pressure. Laser speckle flowgraphy (LSFG) represents a non-invasive method to quantify ocular perfusion also at the ONH. LSFG enables noninvasive quantification of microcirculation of the optic disc in Japanese glaucoma patients.

Study Objectives:

To assess the changes in LSFG parameters in patients with normal tension glaucoma, compared to healthy subjects during flicker light stimulation and isometric exercises.

ELIGIBILITY:
1. Study population: patients with normal tension glaucoma

   * Caucasian men and women aged over 50 years
   * Subject is generally healthy with no current significant or a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination. A significant disorder is defined as a disease or medical condition associated with impaired health status, requiring regular or current medical treatment and/or follow up. For the purposes of this study, an investigator may classify a medical condition as a nonsignificant disorder despite the fact that the subject receives treatment. Subjects having controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90-99 mmHg diastolic) are eligible for participation in this study
   * Normal open angle in a gonioscopic examination
   * Presence of glaucomatous optic disc changes in biomicroscopy and
   * Visual field defects in at least two visual field examinations (Reliability criteria: fixation errors < 20%, false positives < 15%, and false negatives < 33%) Or
   * Abnormal circumpapillary retinal nerve fiber layer thinning (RNFL evaluated by OCT)
2. Control group

   * Men and women aged over 18 years
   * Subject is generally healthy with no current significant or a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination. A significant disorder is defined as a disease or medical condition associated with impaired health status, requiring regular or current medical treatment and/or follow up. For the purposes of this study, an investigator may classify a medical condition as a nonsignificant disorder despite the fact that the subject receives treatment. Subjects having controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90-99 mmHg diastolic) are eligible for participation in this study
   * Baseline IOP in both eyes below 21 mm Hg
   * Normal findings in slitlamp and funduscopic examination

Exclusion Criteria:

* a) Study population: patients with normal tension glaucoma
* History of ocular or systemic disease causing optic nerve damage
* History of IOP greater than 21 mm Hg (corrected by CCT)
* Participation in a clinical trial in the 3 weeks preceding the study
* Ocular surgery (including intravitreal injection) during the 3 months preceding the study
* Ametropia > 6 Dpt
* Smoking
* pre- or perimenopausal women
* Relevant ophthalmic diseases/conditions that could interfere with LSFG measurements (e.g. optic nerve head drusen, tilted disc, etc.)
* Opacities of the cornea (e.g. corneal scars, corneal oedema), the lens (e.g. LOCS-II grading > 2, posterior capsule opacification) or the vitreous (e.g. vitreous haemorrhage, asteroid hyalosis)
* Patients who are not able to cooperate or with insufficient ability to fixate (tremor, nystagmus)
* Blood donation in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ocular infection or clinically significant inflammation
* Pregnancy, planned pregnancy or lactating

  b) Control group
* Abnormal RNFL
* Visual field defects
* Participation in a clinical trial in the 3 weeks preceding the study
* Ocular surgery (including intravitreal injection) during the 3 months preceding the study
* Ametropia > 6 Dpt
* Smoking
* Relevant ophthalmic diseases/conditions that could interfere with LSFG measurements (e.g. optic nerve head drusen, tilted disc, etc.)
* Opacities of the cornea (e.g. corneal scars, corneal oedema), the lens (e.g. LOCS-II grading > 2, posterior capsule opacification) or the vitreous (e.g. vitreous haemorrhage, asteroid hyalosis)
* Patients who are not able to cooperate or with insufficient ability to fixate (tremor, nystagmus)
* Blood donation in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ocular infection or clinically significant inflammation
* Pregnancy, planned pregnancy or lactating

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Change in mean blur rate | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, Prof., Principal Investigator — Allgemeines Krankenhaus Linz
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No